CLINICAL TRIAL: NCT06784453
Title: Evolution of Nutritional Status and Intestinal Function During the Course of the Disease in Patients With Mitochondrial Neurogastrointestinal Encephalomyopathy (Mitochondrial Neurogastrointestinal Encephalomyopathy; MNGIE)
Brief Title: Evolution of Nutritional Status and Intestinal Function in Patients With MNGIE
Acronym: SN-FI_MNGIE
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SN-FI_in_MNGIE
Record Dates: First submitted 2024-11-28; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: Mitochondrial Neurogastrointestinal Encephalopathy Disease
Keywords: Nutritional status in MNGIE; Intestinal function in MNGIE
MeSH Terms: conditions — Visceral myopathy familial external ophthalmoplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort of patients with MNGIE: cohort of patients with MNGIE cared for at the Regional Reference Center for Benign Chronic Intestininal Failure

SUMMARY:
Mitochondrial neurogastrointestinal encephalomyopathy syndrome (MNGIE) is a rare disease characterized by severe gastrointestinal and neurological dysfunction. Its prevalence is 1-9 caIt is a genetic syndrome, with autosomal recessive inheritance, due to mutations in the nuclear gene TYMP (located on chromosome 22q13.32-qter) which encodes the protein thymidine phosphorylase (TP), an enzyme involved in the phosphorylation of the thymidine nucleoside. These mutations result in a significant reduction or complete absence of the enzyme's activity. There is therefore an increase in plasma levels of thymidine and its metabolites, thymidine nucleoside (dThd) and deoxyuridine (dUrd), with toxic accumulation both at a systemic and tissue level, which induces damage and depletion of mitochondrial DNA (mtDNA), multiple deletions and point mutationsses per 1000,000. It is included in the portal of rare diseases and orphan drugs. This syndrome is characterized by severe gastrointestinal and neurological disorders. Gastrointestinal symptoms are the main manifestation of the disease. They are present in 57% of cases at onset and in 100% of cases at diagnosis. Patients present with diarrhea, abdominal pain, borborygmi, vomiting, symptoms of intestinal pseudo-obstruction (32%-65% of cases), weight loss and cachexia (100% of cases). The symptoms, due to the progressive accumulation of metabolites toxic to mitochondrial DNA, are cumulative and evolutionary over time. The available therapeutic options (peritoneal dialysis, platelet infusion and enzyme replacement therapy) are unable to produce lasting clinical improvement. The drastic reduction in weight, resulting from the inability of patients to eat effectively orally, requires the use of home parenteral nutrition (NPD) in almost all cases.

The objective of the study is to describe the evolution of the nutritional status and intestinal function during the course of the disease in patients with MNGIE.

DETAILED DESCRIPTION:
This is a drug-free observational study, both retrospective and prospective, single-center carried out on adult patients with MNGIE, followed at the Regional Reference Center for Benign Chronic Intestinal Insufficiency-Pironi of the IRCCS-AOUBo based on data collected during clinical follow-up at the same centre. The data will be collected in a structured manner using the information present in the medical records obtained in the past as part of normal clinical practice for patients already in the care of the Center at the time of inclusion in the study and that obtained at the time of taking charge of the Center and during clinical follow-up, for new patients.

The study is an observational study without drug and does not involve any study-specific treatment or visit, but exclusively the structured collection of information obtained in the past as part of normal practice (clinical records and related documents) for the retrospective phase and the registration of clinical data collected during the normal care process (follow-up), for the prospective phase. The study does not include any study-specific visits The data will be collected at quarterly intervals starting from the moment the Center takes charge of the patients (time T0).

The following data relating to the history of the disease will also be collected: age at onset of symptoms, age at diagnosis, symptoms and signs at onset, symptoms and signs at diagnosis, symptoms and signs during clinical follow-up. The study population consists of patients with MNGIE followed at the SSD-Clinical Nutrition and Metabolism - Regional Reference Center for Benign Chronic Intestinal Insufficiency-Pironi of the AOU-Policlinico di Sant'Orsola.

MNGIE is a rare syndrome for which a prevalence of 1-9 cases per million inhabitants is described. In Italy there are about ten confirmed cases. To date, the Center has followed 8 patients with MNGIE, of which 6 are currently still in the care of the center and two have died.

It will also be necessary to use the data of patients who did not give consent because they had died or were no longer associated with our center, since failure to involve this population would reduce the eligible sample, producing negative consequences for the study in terms of the significance of the results. Therefore, in the case of deceased or untraceable patients following every reasonable effort made to contact them (via postal address, contact with the general practitioner or via telephone call but only in cases in which the patient had previously expressed consent to telephone contact ), on the basis of General Authorization no. 9 to the processing of personal data carried out for scientific research purposes, issued by the Guarantor on 11/12/2014, the processing of personal data will be carried out in the absence of consent.

For each patient meeting the inclusion criteria, the following parameters will be recorded in a structured way at time T0 (time of taking charge of the patient by the Centre) and at subsequent quarterly intervals:

* Personal data: Age, gender
* Vital parameters: Blood pressure (BP) and heart rate (HR)
* Laboratory tests. Hemoglobin (Hb) and MCV, serum iron (Fe), ferritin, albumin, prealbumin, glycemia, triglycerides, total cholesterol, HDL cholesterol, uric acid, lactic acid, serum bicarbonates, lipase, electrolytes and serum mineral salts (Nas, Ks, Cls, Cas, Ps, Mgs), trace elements (Cu, Zn, Sel), ceruloplasmin, parathyroid hormone (PTH), osteocalcin, cross laps; Urine: chemical-physical examination, electrolytes and urinary mineral salts ([Nau, Ku, Clu, Cau, Pu, Mgu]), thymidine and deoxyuridine dosage;
* Nutrition status. Weight history: healthy weight, weight at diagnosis, current weight), height, body mass index (BMI kg/h (m)2); body composition: with impedance measurement [body cell mass (BCM), fat mass (FM), total water (TBW), extracellular water (ECW), phase angle] and with total body bone densitometry (DEXA) [lean mass (FFM), fat mass (FM)]; bone mineral density (MBD): L1-L4 and femoral neck: MBD (g/cm3), T-score, Z-score; vitamins: folate, vitamin B12, vitamin 25D, vitamin A, vitamin E, vitE/(TGL+Col) ratio; hand grip strength (kg)
* Energy balance: food intake (diary/survey), evaluation of appetite (absent, low, preserved, increased), type of diet (water, liquid, creamy, free of waste and lactose, low-lipid, free); Basal energy expenditure (BEE) calculated according to the Harris-Benedict equation and measured with indirect calorimetry; Total energy expenditure (TEE): calculated (BEEx Physical Activity Level [LAF]) and measured with Sensewear-Armband slide.
* Intestinal absorption: lipid absorption (Wandekamer micromethod), energy absorption (energy absorption % = 100-lipid excretion+10).
* Intestinal protein dispersion: clearance of fecal alpha-1 antitrypsin
* Intestinal motility: bowel characteristics, clinical evaluation and instrumental evaluation through direct abdominal x-ray, gastrointestinal manometry; investigation for the presence of intestinal bacterial hyperproliferation syndrome (SIBO) with breath test-lactulose or glucose and/or; Fecal calprotectin. • Endoscopic investigations: esophagogastroduodenoscopies (EGDS), rectoscopies (RCS)
* Complete abdominal ultrasound with study of the loops and hepatic elastometry
* Nutritional therapies

  * Home Parenteral Nutrition (NPD). Characteristics of the nutritional mixture [volume (mL/day), caloric intake (Kcal/day); bromatological composition (amino acids, carbohydrates, lipids (g/day and Kcal/day), vitamins and trace elements]; number of weekly infusions;
  * Oral nutritional supplements (type and quantity/day)
* Transplant therapy if carried out Marrow transplant or liver transplant (date and clinical progress). The following data relating to the history of the disease will also be collected: age at onset of symptoms, age at diagnosis, symptoms and signs at onset, symptoms and signs at diagnosis, symptoms and signs during clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MNGIE (positive genetic investigation for the presence of mutation of the nuclear TYMP gene).
* Obtaining informed consent

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients with MNGIE followed at the Regional Reference Center for Benign Chronic Intestinal Insufficiency-Pironi of the IRCCS AOUBo
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Nutritional status 1 | at well being, at diagnosis of MNGIE, at FUP every four months, at last FUP/death
  BMI
Nutritional status 2 | at well being, at diagnosis of MNGIE, at FUP every four months, at last FUP/death
  Body composition by bioimpedance analysis when available
Nutritional status 3 | at well being, at diagnosis of MNGIE, at FUP every four months, at last FUP/death
  Serum Albumin (mg/L) when available

CONTACTS AND LOCATIONS:
Overall Officials: Loris Pironi, MD, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy (+39), Italy